CLINICAL TRIAL: NCT00317317
Title: Acupuncture for Infertility Patients: The Effect on IVF
Brief Title: The Effect of Acupuncture on Infertility With In-Vitro Fertilization (IVF) Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Principal Investigator, Grant G. Zhang, Assistant Professor, National Center for Complementary and Integrative Health (NCCIH)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R21AT002651-01A1 (NIH)
Record Dates: First submitted 2006-04-20; First posted 2006-04-24 (Estimated); Last update posted 2019-09-11 (Actual); Status verified 2009-08

CONDITIONS: Infertility
Keywords: IVF; Acupuncture; Pregnant
MeSH Terms: conditions — Infertility | interventions — Acupuncture Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: Acupuncture — 4 acupuncture treatments will be conducted during the IVF cycle. The 1st one is at the beginning of egg stimulation, the 2nd one is before the egg retrieval, the 3rd and 4th one are before and after the embryo transfer

SUMMARY:
Infertility is a common problem with increased incidence. In-vitro fertilization (IVF) is by far the most commonly used treatment. The success rate of IVF is still low. This study examines the effect of acupuncture on IVF pregnancy rate, as well as possible mechanisms. It is hypothesized that acupuncture can significantly increase the IVF pregnancy rate.

DETAILED DESCRIPTION:
Infertility is a common health problem in the United States with approximately 15% of women of childbearing age receiving care for this disorder. One of the most successful and commonly utilized treatment options is in-vitro fertilization (IVF). Data collected by the Center for Disease Control (CDC) and the Society for Assisted Reproduction (SART) showed that in the year 2001, over 100,000 IVF treatment cycles were performed through the more than 400 IVF centers in the U.S. Despite many recent technological advances, pregnancy rates with IVF remain limited with the most recent CDC/SART data reporting that only 27% of treatment cycles result in a live birth. Acupuncture has been utilized in China for centuries to regulate the female reproductive system and has in recent years become a popular option for infertile couples in the States. Though acupuncture has been studied in other infertility settings, IVF is chosen because:

1. IVF is one of the most common infertility treatments as well as the most resource intensive treatment option. Therefore, an improvement in IVF success will provide the greatest benefit to patients and society.
2. IVF affords a unique opportunity to gather the most data regarding the reproductive process and to investigate putative acupuncture related physiological changes.

We propose a randomized, sham controlled feasibility study on the effect of acupuncture on IVF. Sixty IVF patients will be recruited into the study to accomplish the following aims:

1. To examine the feasibility of recruiting and retaining a sufficient number of patients for an adequate powered study,
2. To identify issues related to the multicenter approach that could alter study endpoints,
3. To examine the effect size of the treatment group as compared to the sham group,
4. To examine whether acupuncture is a safe procedure for women undergoing IVF,
5. To examine the effect of acupuncture on clinical IVF outcomes, and
6. To examine the physiological and psychological impact of acupuncture on IVF patients.

Results obtained from the study will provide necessary information for a larger, definitive study, as well as knowledge regarding the broad mechanism of acupuncture on female reproductive function.

ELIGIBILITY:
Inclusion Criteria:

* Patient is undergoing in-vitro fertilization protocol (both IVF and intracytoplasmic sperm injection - ICSI)
* Patient is acupuncture naïve.
* Patient has basal serum follicle-stimulating hormone (FSH) < 10
* Patient has given informed consent to participate in study

Exclusion Criteria:

* Patient has had acupuncture performed previously or currently
* Patient has basal serum FSH of 10 or more

Min Age: 21 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2005-10; Primary Completion 2009-02 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
Clinical pregnancy rate | 6 to 8 weeks

SECONDARY OUTCOMES:
Miscarriage rate | one year
Take home baby rate | one year
B-endorphin levels | 2 weeks
Stress measurement | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Grant Zhang, Ph.D., Principal Investigator — Center For Integrative Medicine, University of Maryland
Locations (2):
- United States (2):
  - Reproductive Endocrinology and Infertility, Dept. of OB/GYN, Baltimore, Maryland
  - The GBMC Fertility Center, Baltimore, Maryland

REFERENCES:
- [Background] Paulus WE, Zhang M, Strehler E, El-Danasouri I, Sterzik K. Influence of acupuncture on the pregnancy rate in patients who undergo assisted reproduction therapy. Fertil Steril. 2002 Apr;77(4):721-4. doi: 10.1016/s0015-0282(01)03273-3. PMID 11937123